CLINICAL TRIAL: NCT03856697
Title: A Randomized Controlled, Double-blind, Multicenter, Phase III Clinical Study to Compare Efficacy and Safety of Abivertinib Maleate Versus First-line Standard Therapy EGFR-TKI in Patients With Advanced NSCLC With Sensitive EGFR Mutation
Brief Title: Abivertinib Maleate Versus Geifitinib in Patients With Advanced Non-small Cell Lung Cancer With Sensitive EGFR Mutation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hangzhou ACEA Pharmaceutical Research Co., Ltd. (Industry)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AC201812AVTN04
Record Dates: First submitted 2019-02-20; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Advanced Non-small Cell Lung Cancer
MeSH Terms: interventions — abivertinib; Gefitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abivertinib Maleate Capsules+ Placebo Gefitinib Tablets (Experimental): Abivertinib Maleate Capsules (300 mg , orally, twice daily) plus Placebo Gefitinib Tablets (250 mg orally, once daily), in accordance with the randomization schedule.
  Interventions: Drug: Abivertinib Maleate Capsules; Drug: Placebo Gefitinib Tablets
- Gefitinib Tablets+ Placebo Abivertinib Maleate Capsules (Active Comparator): Placebo Abivertinib Maleate Capsules (300 mg , orally, twice daily) plus Gefitinib Tablets(250 mg orally, once daily), in accordance with the randomization schedule.
  Interventions: Drug: Gefitinib Tablets; Drug: Placebo Abivertinib Maleate Capsules

INTERVENTIONS:
Drug: Abivertinib Maleate Capsules — patients receive the test drug (Abivertinib maleate Capsules) since the first day of cycle 1. One cycle is defined as 21 days. The patient shall take the study drugs twice a day. The first dose is 3 capsules, and the second dose is 3 capsules. The drugs should be administered with water before or after meals.
  Arms: Abivertinib Maleate Capsules+ Placebo Gefitinib Tablets
Drug: Placebo Gefitinib Tablets — patients receive the test drug (Placebo Gefitinib Tablets) since the first day of cycle 1. One cycle is defined as 21 days. The patient shall take the study drugs twice a day. The first dose is 1 tablet. The drugs should be administered with water before or after meals.
  Arms: Abivertinib Maleate Capsules+ Placebo Gefitinib Tablets
Drug: Gefitinib Tablets — patients receive the control drug (Gefitinib Tablets) since the first day of cycle 1. One cycle is defined as 21 days. The patient shall take the study drugs twice a day. The first dose is 1 tablet. The drugs should be administered with water before or after meals.
  Arms: Gefitinib Tablets+ Placebo Abivertinib Maleate Capsules
Drug: Placebo Abivertinib Maleate Capsules — patients receive the control drug (Placebo Abivertinib Maleate Capsules) since the first day of cycle 1. One cycle is defined as 21 days. The patient shall take the study drugs twice a day. The first dose is 3 capsules, and the second dose is 3 capsules. The drugs should be administered with water before or after meals.
  Arms: Gefitinib Tablets+ Placebo Abivertinib Maleate Capsules

SUMMARY:
To compare efficacy and safety of Abivertinib maleate alone versus standard first-line EGFR-TKIs for the treatment of patients with advanced non-small cell lung cancer with sensitive EGFR mutation

DETAILED DESCRIPTION:
This is a randomized controlled, double-blind, multicenter, phase III clinical study to compare efficacy and safety of Abivertinib maleate versus first-line standard therapy EGFR-TKI for the treatment of patients with advanced non-small cell lung cancer with sensitive EGFR mutation

ELIGIBILITY:
Inclusion Criteria:

1. Stage IV NSCLC confirmed by histology or cytology, or Stage IIIB-IIIC stage NSCLC not suitable for radical surgery or radiation therapy (eighth edition lung cancer staging criteria of International Association for the Study of Lung Cancer).
2. At least one lesion that can be measured by imaging examinations (CT, MRI) according to Response Evaluation Criteria in Solid Tumors (RECIST) V1.1; the lesion can be accurately and reproducibly measured at baseline. Long diameter of tumor in CT and MRI scan ≥ 10mm, or short diameter of metastatic lymph node ≥15 mm, and the lesion has not undergone radiotherapy or biopsy (if the patient has only one target lesion and requires biopsy, biopsy of the target lesion is allowed, but time interval between biopsy and baseline assessment of tumor during screening period must be ≥2 weeks, and the target lesion after biopsy still meets the definition of target lesion per RECIST); the lesion either has no radiotherapy history or no obvious disease progression after radiotherapy.
3. Patients with or without brain metastases could be enrolled. For patients with symptomatic brain metastases, brain lesions must be stable, and the patients shall not receive hormonal therapy within 2 weeks before start of the study treatment. In addition, the Investigator shall confirm that local treatment for the brain metastases is temporarily not needed, and PS score does not decrease significantly in the last 2 weeks. If the patient has received brain radiotherapy, time interval between end of radiotherapy and start of the study treatment shall exceed 2 weeks, and radiotherapy-related toxicity shall be recovered to less than or equal to grade 1 (CTCAE criteria) (except for hair loss)Investigator.
4. Tumor tissue or cytopathological specimens have any of two common sensitive EGFR mutation (Ex19del or L858R) as confirmed by tests with Cobas (Roche) kit in central lab of this study, which can be combined with other EGFR gene mutations.
5. The patients shall have sufficient vital organ functions during screening, including:

   * Absolute neutrophil count (ANC) ≥ 1.5x10^9/L if no treatment with hematopoietic stimulating factor is performed within 14 days before the first dose
   * Platelet count ≥100×10^9/L if no treatment with hematopoietic stimulating factor or blood transfusion is performed within 14 days before the first dose
   * Hemoglobin >90g/L if no treatment with hematopoietic stimulating factor or blood transfusion is performed within 14 days before the first dose
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5X ULN (ULN = upper limit of normal) for patients without liver metastasis, or aspartate aminotransferase (AST), alanine Acid transaminase (ALT) ≤ 5 X ULN (ULN = upper limit of normal) for patients with liver metastasis
   * Total bilirubin ≤1.5X ULN
   * Coagulation function INR ≤ 1.5
   * Serum creatinine ≤ 1.5 × ULN or creatinine clearance rate (calculated using the Cockcroft and Gault formula) ≥ 50 ml/min
6. Palliative radiotherapy is allowed to be completed before 1 week prior to study enrollment, and radiotherapy-related toxicity shall be recovered to less than or equal to grade 1 (CTCAE 5.0).
7. ECOG score: 0 or 1 point, and no signs of deterioration should be found in the last 2 weeks; expected survival time >12 weeks.
8. Negative results in pregnancy tests (only for women with fertility potential). No fertility potential is defined as at least 1 year after menopause or surgical sterilization or hysterectomy.
9. All enrolled patients (whether male or female) agree to take effective contraceptive measures throughout the treatment period and at least 3 months after the end of treatment.

   For women with fertility potential, effective contraceptive methods include:

   Any combination of the following two methods (a+b or a+c or b+c):
   1. Use of oral, injection or implantable hormonal contraceptive methods or other forms of hormonal contraception with similar efficiency (failure rate ≤ 1%), such as hormone vaginal ring or percutaneous hormonal contraception
   2. implantation of intrauterine device (IUD) or intrauterine system (IUS)
   3. Barrier contraception method: a condom or a cervical cap (diaphragm or cervical cap) coated with spermicidal foam/gel/cream/vaginal suppository Note: Complete abstinence (if it is the patient's preferred and usual lifestyle), periodic abstinence (such as calendar method, ovulation method, symptomatic temperature method and post-ovulation method) and in vitro ejaculation are unacceptable methods of contraception.

   If a woman has at least 12 months of natural amenorrhea and meets the clinical criteria for postmenopausal woman or has undergone bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 weeks ago, she is considered a postmenopausal woman and does not have fertility potential.

   Men who have sex shall use condoms during sexual intercourse during the medication and within 3 months after end of treatment, so as not to conceive their sexual partners.

   Men who have vasectomy shall also use condoms to prevent the transmission of drugs through semen.
10. Patients shall voluntarily participate in the study, sign the informed consent form, follow the study treatment plan and visit plan, and be able to cooperate in observation of adverse events and efficacy

Exclusion Criteria:

1. History of systemic chemotherapy or any other systemic treatment for advanced NSCLC, including:

   * Systematic chemotherapy, biotherapy, immunotherapy or any study drug treatment (patients who have previously received preoperative neoadjuvant chemotherapy or postoperative adjuvant chemotherapy or radical chemoradiotherapy can be enrolled if disease progression occurs after one year following the last treatment)
   * Any EGFR TKI drug
   * Any anti-tumor Chinese medicine (the patients who have received no more than 3 doses (1 dose per administration) of Chinese medicine with anti-tumor effects can be enrolled, but the medicine shall be discontinued for at least 2 weeks before treatment with the study drug)
2. The patients who are currently receiving a known strong cytochrome P450 (CYP)3A4 inhibitor or inducer (or the patients who cannot discontinue the drug within 1 week prior to the first dose of study drug);
3. Acute and chronic hepatitis C, HBsAg positive and/or HBV DNA positive;
4. HIV antibody positive, or other acquired, congenital immunodeficiency disease, or a history of organ transplantation;
5. A history of interstitial lung disease, or clinically significant radiation pneumonitis or imaging findings suggesting interstitial pneumonia or radiation pneumonitis;
6. Evidence of severe or uncontrolled systemic diseases (such as severe mental disease, neurological diseases, epilepsy or dementia, unstable or uncompensated diseases in respiratory, cardiovascular, liver, or kidney, uncontrolled hypertension [ CTCAE grade 2 above hypertension after drug treatment];
7. Patients with active bleeding or thrombotic disease who are taking therapeutic anticoagulant drugs or have bleeding tendency.
8. There are clinically significant abnormalities in rhythm, conduction and morphology in resting electrocardiogram, such as complete left bundle branch block, heart block above grade II and PR interval >250 ms; myocardial infarction in the past 6 months; risk factors leading to prolongation of QT interval or increasing risk factors for arrhythmia, such as heart failure, hypokalemia (greater than or equal to CTCAE grade 2), confirmed or suspected congenital long QT syndrome, family history of long QT syndrome or history of sudden death under 40 years old of first-degree relatives; mean QT interval (QTcB) after correction of Bazetts of 3 ECGs: male > 450 milliseconds, female > 470 milliseconds.
9. The Investigator's concerns based on safety or compliance with clinical study process, or conditions that may interfere with interpretation of study results, including but not limited to: active infections/inflammations and any other serious and unstable diseases, intestinal obstruction, inability to swallow drugs, social/psychological issues, etc.
10. In addition to NSCLC, another malignant disease has been diagnosed in the past 5 years (excluding malignant tumors that have been cured, such as completely excised basal cell carcinoma, carcinoma in situ, and thyroid cancer).
11. Patients underwent extensive bone marrow radiation therapy within 4 weeks prior to use of the study drug.
12. Surgery was performed ≤ 28 days before use of the study drug (except for surgery for biopsy).
13. Use of any drugs known to prolong QT interval or incapability to stop using these drugs within 2 weeks before the first dose of study drug;
14. Use of immunosuppressive therapy within 1 month before initiation of study treatment;
15. Patients with previous treatment with this study drug or known to be allergic to the study drug ingredients or excipients cannot be enrolled;
16. Patients who withdrew from the study cannot be enrolled.
17. Pregnant or lactating women;
18. Other potential risks based on which the Investigator believes that the patients are not suitable for participating in this study.
19. Gastrointestinal perforation and/or Keratitis history within 1 year before initiation of study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Assess the efficacy of Abivertinib: Progression Free Survival (PFS) | From baseline, then every 6 weeks, until disease progression or discontinuation from study. From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Progression-free survival (PFS) of Abivertinib maleate alone versus standard first-line EGFR-TKI for the treatment of treatment-naïve patients with advanced non-small cell lung cancer with sensitive EGFR mutation (Investigator's evaluation according to RECIST1.1 criteria)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | At baseline and every 6 weeks until the date of first documented progression or date of death from any cause ( approximately 12 months)
  Objective Response Rate (ORR) of Abivertinib maleate alone versus standard first-line EGFR-TKI for the treatment of treatment-naïve patients with advanced non-small cell lung cancer with sensitive EGFR mutation
Disease Control Rate (DCR) | At baseline and every 6 weeks until the date of first documented progression or date of death from any cause ( approximately 12 months)
  Disease Control Rate (DCR) of Abivertinib maleate alone versus standard first-line EGFR-TKI for the treatment of treatment-naïve patients with advanced non-small cell lung cancer with sensitive EGFR mutation
Duration of Response (DoR) | At baseline and every 6 weeks until the date of first documented progression or date of death from any cause ( approximately 12 months)
  Duration of Response (DoR) of Abivertinib maleate alone versus standard first-line EGFR-TKI for the treatment of treatment-naïve patients with advanced non-small cell lung cancer with sensitive EGFR mutation
Overall Survival (OS) | From first dose to end of study or date of death from any cause, whichever comes first, assessed every 6 weeks (approximately 36 months)
  Overall Survival (OS) of Abivertinib maleate alone versus standard first-line EGFR-TKI for the treatment of treatment-naïve patients with advanced non-small cell lung cancer with sensitive EGFR mutation
Safety and Resistance: Number and severity of AEs/SAEs | From screening to the end of survival follow-up, which is assessed through study completion until 30 days after discontinuation
  Number and severity of AEs/SAEs of Abivertinib maleate alone versus standard first-line EGFR-TKI for the treatment of treatment-naïve patients with advanced non-small cell lung cancer with sensitive EGFR mutation
Safety and Resistance: Drug exposure | Continuously throughout the study until 30days after discontinuation
  The mean, standard deviation, maximum, minimum, and median of drug exposures in the two groups are described
Safety and Resistance: General physical examination status | Continuously throughout the study until 30days after discontinuation
  A general physical examination includes: general status, skin, head and neck (includes: eyes, ears, nose, throat), respiratory system, cardiovascular system, abdomen,superficial lymph nodes, thyroid, musculoskeletal system (including spine and limbs), and nervous system, and any other physical signs of clinical significance. During the treatment, physical examination of the potentially affected organs will be performed.
Safety and Resistance: Electrocardiogram(ECG test) | Continuously throughout the study until 30days after discontinuation
  Descriptive statistical analysis of clinical diagnosis results of ECG examination and changes compared with baseline are performed at planned time points, and abnormal ECG examination results are listed.
Safety and Resistance: Eastern Clinical Oncology Group Scores | Continuously throughout the study until 30days after discontinuation
  ECOG (Eastern Clinical Oncology Group) Performance Status Grading Criteria: Range from 0-5, 0 considered to be the best outcome and 5 to be the worst outcome
Questionnaire: Health-related quality of life (HRQoL) | At baseline and every 6 weeks until the date of first documented progression or date of death from any cause ( approximately 12 months)
  Quality of life questionnaire of Abivertinib maleate alone versus standard which includes 5 functional domains, 3 symptom domains, 1 overall health status/quality of life domain and 6 single entries. Standardized scores of the domains/single entries in the questionnaire are used to statistically describe the absolute values and changes from baseline at each evaluation time point; t test is used to compare changes from baseline in overall quality of life score at each evaluation time point in both groups; analysis of variance is used to compare changes in overall health status score at each evaluation time point between the two groups. first-line EGFR-TKI for the treatment of treatment-naïve patients with advanced non-small cell lung cancer with sensitive EGFR mutation

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provicial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No